CLINICAL TRIAL: NCT05591378
Title: Comparison of Core Stability and Otago Exercise on Balance and Quality of Life in Patients With Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: abdul mansoor
Record Dates: First submitted 2022-09-21; First posted 2022-10-24 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Stroke
Keywords: balance; quality of life; stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- core stability exercises (Experimental): improve balance and muscle strengthening
  Interventions: Other: core stability exercises
- otago exercises (Experimental): improve balance and quality of life
  Interventions: Other: otago exercises

INTERVENTIONS:
Other: core stability exercises — exercises for 8 weeks and 3 individual sessions per week for 30-45 minutes. Each exercise will be given for 3 to 5 minuts.
  first week:Cat camel stretch, all fours stretch and lifting one leg, cobra pose, lying on your back and raising the legs/one leg, and hamstring stretch on chair second week:Straight Leg Crunch, with first week exercises third week:Crunch, bridge exercise,and lifting the legs/one leg straight out with first week exercises fourth week:lifting the legs/one leg to the opposite hand, with first week exercises fifth week:Reverse Crunch, bridge exercise without support with first week exercises sixth week:Hamstring stretch on the Floor with first week exercises seventh week:lifting one hand and one leg, with first week exercises eight week:Exercise Ball Crunch,and stability ball bridge with first week exercise
  Arms: core stability exercises
Other: otago exercises — exercises for 8 weeks and 3 individual sessions per week for 30-45 minutes. Each exercise will be given for 3 to 5 minuts.
  Walking forward with support, standing on heel with support, side walking with support, standing on one foot with support.Walking forward without support, standing on heel without support, side walking without support, standing on one foot without support.
  Walking backward with support, walking on heel with support, walking and turning around, walking on heel with support.
  Walking backward without support, walking on heel without support, walking and turning around, walking on heel without
  Arms: otago exercises

SUMMARY:
Core stability and otago exercise program has been proved to be effective in many conditions like muscles strenghing, gait improvement and relieving of pain. Hence the aim of present study is to compare the effectivness of Core stability and Otago exercise on balance and quality of life in patients with stroke.

DETAILED DESCRIPTION:
The Otago Exercise Program (OEP), consist of resistance training and balance training exercises. The OEP is composed of three domains, namely muscle strengthening, balance training with a progression by increasing ankle cuff weights and number of sets, in association with a walking plan. It is a program that incorporates moderate intensity strength exercises focusing on the lower limbs and balance to be performed for about 30 min at least three times a weekStrength training consisted of flexion and extension exercises of the knee, ankle, and toe joints, as well as hip opening exercises to strengthen the sides of the pelvis. Balance training consisted of walking backwards, walking in a figure of eight, heel-toe walking, standing on one leg, walking on the heels, walking on the toes, heel-toe walking backwards, standing up from a sitting position, and walking up stairs.exercises and physical activities could promote balance, flexibility, muscular strength, and walking ability among elderly people.OEP three times a week, for 6 months, can improve dynamic balance.core stability exercises for five weeks in addition to conventional physiotherapy five days a week for the same period, improved dynamic sitting balance, standing balance, gait and activities of daily living at the post intervention assessment in subacute post-stroke survivors.

ELIGIBILITY:
Inclusion Criteria:

* Sub acute stroke(3 to 6 months).
* Ashworth scale 1 to 3.
* Patients having cognition level is (26-30) according to MOCA.
* Patients having (21 to 42) score according to BBS.

Exclusion Criteria:

* Fractures.
* Participants with recurrent stroke.
* Participants with sever spasticity
* Orthopedic or other neurological impairment that could influence balance.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2022-11-20 (Actual); Primary Completion 2023-04-15 (Actual); Study Completion 2023-04-15 (Actual)

PRIMARY OUTCOMES:
Berg balance scale | 8 week
  The Berg Balance Scale (BBS) is used to objectively determine a patient's ability (or inability) to safely balance during a series of predetermined tasks. It is a 14 item list with each item consisting of a five-point ordinal scale ranging from 0 to 4, with 0 indicating the lowest level of function and 4 the highest level of function.

SECONDARY OUTCOMES:
Functional independence measure | 8 week
  Functional independence measure scale is used to measures of independence for self-care.
  Functional independence measure scale assess six area of function including sphincter control, transfers, locomotion, communication, and social cognition. Each item is scored on a 7 point ordinal scale, ranging from a score of 1 to a score of 7. The higher the score, the more independent the patient is in performing the task associated with that item.
Stroke specific quality of life questionnaire | 8 week
  Specific Quality Of Life scale is a patient-centered outcome measure intended to provide an assessment of health-related quality of life specific to patients with stroke.

CONTACTS AND LOCATIONS:
Overall Officials: sania aziz, MSNMPT, Principal Investigator — Riphah International University
Locations (1):
- Bacha khan medical complex, Swābi, Kpk, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chung EJ, Kim JH, Lee BH. The effects of core stabilization exercise on dynamic balance and gait function in stroke patients. J Phys Ther Sci. 2013 Jul;25(7):803-6. doi: 10.1589/jpts.25.803. Epub 2013 Aug 20. PMID 24259857
- [Background] Cabanas-Valdes R, Bagur-Calafat C, Girabent-Farres M, Caballero-Gomez FM, Hernandez-Valino M, Urrutia Cuchi G. The effect of additional core stability exercises on improving dynamic sitting balance and trunk control for subacute stroke patients: a randomized controlled trial. Clin Rehabil. 2016 Oct;30(10):1024-1033. doi: 10.1177/0269215515609414. Epub 2015 Oct 8. PMID 26451007
- [Background] Cabanas-Valdes R, Bagur-Calafat C, Girabent-Farres M, Caballero-Gomez FM, du Port de Pontcharra-Serra H, German-Romero A, Urrutia G. Long-term follow-up of a randomized controlled trial on additional core stability exercises training for improving dynamic sitting balance and trunk control in stroke patients. Clin Rehabil. 2017 Nov;31(11):1492-1499. doi: 10.1177/0269215517701804. Epub 2017 Mar 29. PMID 28351168
- [Background] Chiu HL, Yeh TT, Lo YT, Liang PJ, Lee SC. The effects of the Otago Exercise Programme on actual and perceived balance in older adults: A meta-analysis. PLoS One. 2021 Aug 6;16(8):e0255780. doi: 10.1371/journal.pone.0255780. eCollection 2021. PMID 34358276
- [Background] Liu-Ambrose T, Donaldson MG, Ahamed Y, Graf P, Cook WL, Close J, Lord SR, Khan KM. Otago home-based strength and balance retraining improves executive functioning in older fallers: a randomized controlled trial. J Am Geriatr Soc. 2008 Oct;56(10):1821-30. doi: 10.1111/j.1532-5415.2008.01931.x. Epub 2008 Sep 15. PMID 18795987